CLINICAL TRIAL: NCT05472688
Title: My Baby Biome: Infant Stool Samples for Microbiome Health (MBB)
Status: Active, not recruiting | Type: Observational
Sponsor: Persephone Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-2022-01
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — We will be collecting infant fecal samples that we will be retaining. We will only be processing microbial DNA found in the fecal samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
My Baby Biome is an observational study that will use 600 infant stool samples to determine the biomarkers associated with a healthy infant gut. Biomarkers identified in this study will be used to develop precision probiotics and LBPs for improving infant gut health outcomes to the benefit of all infants. Parents will be asked to submit follow-up questionnaires regarding infant immune health to improve insights obtained from the data.

ELIGIBILITY:
Exclusion Criteria:

* Infants under 2 weeks or over 2 months old
* Infants given any antibiotic or probiotic treatments
* Infants delivered prematurely or admitted to the NICU outside of establishment of normal feeding
* Infants with mothers under the age of 18
* Infants with mothers known to have HIV, Hepatitis A, Hepatitis B, Hepatitis C, or SARS-CoV2

Ages: 0 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: It is anticipated that 600 infants will enroll in this study. It is preferred that enrollment is balanced by sex; however, it is not required. All efforts will be made to provide racial/ethnic balance, with a goal of 20% African American and 10% each of patients with Asian or Hispanic descent. Additionally, we will look to maintain a demographic that represents different birth and feeding modes.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the composition of a healthy infant microbiome | 6-12 Months
  Stool samples will be analyzed for bacterial metagenomics, metabolomics, proteomics, and transcriptomics to define biomarkers (such as bacteria or proteins) that are correlated with healthy infants as defined by the accompanying questionnaire.

SECONDARY OUTCOMES:
Evaluate impact of the microbiome on immune adverse events | 7 Years
  Metadata from questionnaires regarding child immune health will be correlated with the metagenomic gut microbiome composition obtained from the stool sample to define the impact of individual strains on immune adverse events (i.e. allergies, diabetes, asthma, eczema)
Build a library of samples and data for future research | 6-12 Months
  Samples will be stored and data saved in a HIPAA-compliant database. Samples will be linked to patient metadata.

CONTACTS AND LOCATIONS:
Locations (1):
- Persephone Biosciences, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Persephone Biosciences Website — https://www.persephonebiosciences.com/clinical-studies/